CLINICAL TRIAL: NCT00284401
Title: Prosthetic Component Relationship of the Reversed Delta III Total Shoulder Prosthesis in the Transverse Plane of the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/102
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Shoulder Prosthesis
Keywords: Reversed prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Evaluation of the placement of the Delta prosthesis

SUMMARY:
Comparison of the function and mobility of the shoulder with the placement of the Delta prosthesis (anteversion and retroversion of the glenoidal and humeral components)

ELIGIBILITY:
Inclusion Criteria:

* Shoulder prosthesis

Exclusion Criteria:

* Inability to place the hand on the back in prone position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-02; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Function and mobility of the shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be